CLINICAL TRIAL: NCT03342586
Title: Changes in Resting State Functional Connectivity in Patients With Central Nervous System Lymphoma Receiving High Dose Chemotherapy and Autologous Stem Cell Transplant
Brief Title: Using a Novel Functional MRI Technique to Evaluate for Neurotoxicity
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-403
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Central Nervous System Lymphoma
Keywords: resting state functional Magnetic Resonance Imaging; rsfMRI; 17-403

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Central Nervous System Lymphoma: Participants will have non-Hodgkins lymphoma involving the brain (primary or secondary)
  Interventions: Diagnostic Test: Resting State fMRI (rsfMRI); Other: Auditory Attention and Executive Functions Test; Other: Memory Test; Other: Motor Speed Test; Other: Self Reported Quality of Life Questionnaire

INTERVENTIONS:
Diagnostic Test: Resting State fMRI (rsfMRI) — rsfMRI before receiving High-dose chemotherapy with autologous stem cell transplantation/HDC-ASCT (pre-HDC-ASCT), at approximately 3 months (+/- 2 weeks) after HDC-ASCT (early post-HDC-ASCT) and approximately 6months (+/- 2 weeks) after HDC-ASCT (late post-HDC-ASCT).
Other: Auditory Attention and Executive Functions Test — * Trail Making Test (Parts A & B): Part A is a timed test of visual scanning and graphomotor speed; AT: 3 minutes. Part B is a timed measure of set-shifting; Administration Time (AT): 5 minutes. Test-retest reliabilities=0.64-0.94.
  * Brief Test of Attention-BTA assesses auditory working memory; AT: 10 minutes. Test-re-test reliability=0.70.
  * Controlled Oral Word Association Test-COWAT is a timed measure of phonemic verbal fluency. It requires the subject to generate as many words as possible, beginning with a given letter of the alphabet (i.e., F, A, and S). The subject is allowed 60 seconds per letter, and the resultant score is the total number of words produced. Test-retest reliability=0.88. AT: 5 minutes.
Other: Memory Test — The Hopkins Verbal Learning Test-Revised (HVLT-R): The HVLT-R is a test of verbal learning and memory.
Other: Motor Speed Test — Grooved Pegboard Test (GPT)-Dominant Hand and Non-Dominant Hand. It is a timed test of manual dexterity, in which the time to completion is scored separately for each hand.
Other: Self Reported Quality of Life Questionnaire — The Functional Assessment of Cancer Therapy-Brain Cancer (FACT-BR Version 4) consists of 46 questions with five domains assessing physical well-being, social/family well-being, emotional well-being, functional well being, additional concerns. The neuropsychological and QOL assessments will be performed by a neuropsychologist or by a trained RSA under the neuropsychologist's direct supervision.

SUMMARY:
The purpose of this study is to test resting state functional Magnetic Resonance Imaging (rsfMRI) scans to see if rsfMRI scans are better than the standard task based fMRI scans at diagnosing or monitoring central nervous system lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent patients with newly diagnosed or recurrent non-Hodgkins lymphoma involving the brain (primary or secondary), as demonstrated by MRI and histologic confirmation either by positive CSF cytology for lymphoma or a monoclonal lymphocyte population defined by cell surface markers, vitreous or uvea biopsy or brain biopsy
* Age 18-80 years
* Treatment plan for HDC-ASCT
* Fluent in English
* Patients who in the judgment of the investigators and/or consenting professional, are able to understand the purpose of the study and provide informed consent will be included.

Exclusion Criteria:

* Claustrophobia
* Any contraindication to the use of contrast and/or general guidelines for MR imaging as per standard Department of Radiology imaging guidelines
* Unable to cooperate for MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, listed protocol investigators, or Neuroradiology research team at Memorial Sloan Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Change in resting state brain networks over time in participants with central nervous system lymphoma before and after treatment with high-dose chemotherapy with autologous stem cell transplantation through resting state fMRI results | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Behroze Vachha, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.mskcc.org